CLINICAL TRIAL: NCT07116109
Title: Neuromodulation + Prolonged Exposure Therapy: Evaluation of a Technology-Enhanced, Entirely Remote 2-Week Integrated Treatment for Pain and PTSD
Brief Title: Neuromodulation + Prolonged Exposure Therapy: Evaluation of a Technology-Enhanced, Integrated Treatment for Pain and PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Melba Hernandez-Tejada, PhD, DHA, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-25-0436
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain; Post Traumatic Stress Disorder (PTSD)
Keywords: PTSD; transcranial Direct Current Stimulation (tDCS); Traumatic Brain Injury (TBI)
MeSH Terms: conditions — Chronic Pain; Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Transcranial Direct Current Stimulation (tDCS) and Massed-Prolonged Exposure (PE) (Experimental)
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Massed-Prolonged Exposure (PE)
- Sham Transcranial Direct Current Stimulation (tDCS) and Massed-Prolonged Exposure (PE) (Sham Comparator)
  Interventions: Behavioral: Massed-Prolonged Exposure (PE); Device: Sham Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — A constant current intensity of 2 Ma electrical current will be administered for 20 min per session/ 10 sessions total daily for 2 weeks (Monday to Friday)using the headgear M1-SO montage placement.
  Arms: Transcranial Direct Current Stimulation (tDCS) and Massed-Prolonged Exposure (PE)
Behavioral: Massed-Prolonged Exposure (PE) — PE will include a) psychoeducation about the common reactions to traumatic events and presentation of the treatment rationale (sessions 1 and 2), b) repeated in vivo exposure to traumatic stimuli (in vivo exercises are assigned as homework during sessions 3 through 10), c) repeated, prolonged, imaginal exposure to traumatic memories (sessions 3 through 10). All sessions will be delivered via telehealth.
Device: Sham Transcranial Direct Current Stimulation (tDCS) — Sham tDCS delivers an active stimulation of 2 Ma electrical current) for a few seconds to mimic the sensations of active tDCS
  Arms: Sham Transcranial Direct Current Stimulation (tDCS) and Massed-Prolonged Exposure (PE)

SUMMARY:
The purpose of this study is to examine comparative effectiveness of two home-based telemedicine delivered interventions: transcranial Direct Current Stimulation (tDCS) combined with Massed Prolonged Exposure (Massed-PE) vs. Sham tDCS combined with Massed PE, focusing on pain and PTSD outcomes, to determine the comparative effectiveness of the two interventions on process outcomes of patient satisfaction, treatment attrition, and treatment compliance and to explore changes in blood biomarkers associated with stress and inflammatory processes related to pain and PTSD symptom improvements following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of musculoskeletal, chronic, non-cancer pain with a rating of ≥ 3 out of 10 on a 0-10 on the Defense and Veterans Pain Rating Scale (DVPRS) and a pain intensity and interference score of 1 standard deviation above PROMIS normative data (see Measures section below). Symptoms will be required to be of at least six months duration and verified diagnosis in their medical chart authorized by informed consent
* Diagnosis of PTSD assigned on the basis of the Clinician Administered PTSD Scale (CAPS-5) and PCL-5 ≥ 30
* willing to participate in study randomization, treatment assignment, and assessments.

Exclusion Criteria:

* Having a household member who is already enrolled in the study
* Active psychosis or dementia at screening
* Suicidal ideation with clear intent
* Current substance dependence
* current opioid medication for pain and/or current use of sodium channel blockers, calcium channel blockers, or N-Methyl-D-aspartate receptor antagonists, because these medications can block tDCS effects
* pregnancy and/or lactation
* concurrent enrollment in another pain clinical trial
* tDCS or medical related contraindications such as open-injury TBI (penetrating injury), seizure disorder (independently of the type of TBI or condition causing the seizure disorder), pregnancy, implanted metal, claustrophobia
* having pain that is not chronic, presence of severe and frequent migraines, fibromyalgia, or pain caused by a primary condition such as cancer.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2029-01-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity as measured by the Defense and Veterans Pain Rating Scale (DVPRS) | Baseline, midpoint(before session 6), post treatment (after session 10) 3 months, 6 months
  The DVPRS is a validated 11-point numeric rating scale and is scored from 0(no pain at all) to 10(worst pain ever possible), higher scores indicate greater pain severity.
Change in PTSD symptoms as assessed by the Clinician-Administered PTSD Scale 5 (CAPS-5) | Baseline, post treatment (after session 10) 3 months, 6 months
  The CAPS-5 is a 30-item structured clinical interview used to assess the presence and severity of Posttraumatic Stress Disorder (PTSD) symptoms according to Diagnostic and Statistical Manual of Mental Disorders(DSM-5)diagnostic criteria. The scale includes 20 core PTSD symptom items rated on a 5-point scale (0-4) for both frequency and intensity. Each item receives a severity score ranging from 0 (absent) to 4 (extreme/incapacitating), for a total score range of 0 to 80. Higher scores indicate greater PTSD symptom severity.

SECONDARY OUTCOMES:
Change in pain intensity as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain 3a Intensity Scale | Baseline, midpoint(before session 6), post treatment (after session 10) 3 months, 6 months
  This is a 3 item questionnaire and each is scored from 1 (no pain) to 5 (very severe) , maximum score of 15. Higher score indicates greater pain intensity
Change in pain interference as assessed by the PROMIS Pain 8a Interference Scale | Baseline, midpoint(before session 6), post treatment (after session 10) 3 months, 6 months
  This is a 8 item questionnaire scored from 1 (not at all) to 5 (very much) , raw score range is 8-40, higher scores indicating greater pain interference.
Change in symptoms of Post-Traumatic Stress Disorder (PTSD)as assessed by the PTSD Checklist-5 Civilian (PCL-5) | Baseline, midpoint(before session 6), post treatment (after session 10) 3 months, 6 months
  This is a 20 item questionnaire each scored from 0(not at all) to 4( extremely), for a total score range of 0-80 higher scores indicating worse outcome
Change in Quality of life as assessed by the World Health Organization Quality of Life - Short Form (WHOQOL-BREF) | Baseline, midpoint(before session 6), post treatment (after session 10) 3 months, 6 months
  This is a 26-item measure categorized into four domains (i.e., physical health, psychological well- being, social relationships, and environment).Each item is rated on a 5-point Likert scale ranging from 1 (low perception) to 5 (high perception). Domain scores are calculated and transformed to a 0-100 scale, with higher scores indicating better perceived quality of life. Two additional items assess overall quality of life and general health.
Change in anxiety as assessed by the Generalized Anxiety Disorder Scale 7 (GAD-7) | Baseline,post treatment (after session 10) 3 months, 6 months
  This is a 7 item questionnaire , each scored from 0( not at all) to 3(nearly every day) for a maximum score range of 0-21 higher scores indicating more anxiety
Quality of sleep as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, post treatment (after session 10) 3 months, 6 months
  The PSQI is a 19-item self-report questionnaire. There are 7 component scores (subjective sleep quality, sleep latency, duration, efficiency, disturbances, medication use, daytime dysfunction) and each is scored from 0 (No difficulty or very good sleep) to 3 ( Severe difficulty) for a score range of 0-21 higher score indicating poor sleep
Change in depression as assessed by the The Patient Health Questionnaire (PHQ-9) | Baseline, post treatment (after session 10) 3 months, 6 months
  This is a 9 item questionnaire and each is scored on a 4 point likert scale from 0(not at all) to 3(nearly every day) for a score range of 0-27 higher scores indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Melba Hernandez-Tejada, PhD, DHA, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No